CLINICAL TRIAL: NCT03397953
Title: Phase II Study of Vinorelbine for Children With Recurrent Anaplastic Large Cell Lymphoma
Brief Title: Vinorelbine for Recurrent ACLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Cancer Group, China (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCGChina-ALCL-ABANDONED
Record Dates: First submitted 2018-01-06; First posted 2018-01-12 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Anaplastic Large Cell Lymphoma; Vinorelbine
Keywords: Anaplastic Large Cell Lymphoma; Childhood; Adolescent; Recurrent; Treatment
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic; Recurrence | interventions — Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vinorelbine monotherapy treatment (Experimental): Patients will be treated by Vinorelbine. Four weeks as a course. There are 20 courses in total.
  Interventions: Drug: Vinorelbine

INTERVENTIONS:
Drug: Vinorelbine — Vinorelbine will be used 25mg/m2/week, rest for 1 week after 3 weeks of continuous use, 4 weeks will be a course. After 1 week there will be a simple assessment, after 2 weeks will be a comprehensive assessment. If the patient got disease progression or partial response/stable disease, he/she would be removed from this trial.

SUMMARY:
The purpose of this study is to assess the efficiency and safety of vinorelbine in the treatment of relapsed / advanced ALCL in children and adolescents.

DETAILED DESCRIPTION:
Anaplastic large cell lymphoma (ALCL) is a rare non-Hodgkin's lymphoma, around 30% patients would get relapse. Vinorelbine(Navelbine) is a third-line treatment option for Hodgkin's disease(HD) after transplantation failed, while both HD and ALCL express CD30. When ALCL recurred, vinblastine monotherapy was used and the 5-year EFS up to 30%, 5-year OS up to 60%. In China vinblastine is unavailable. Vinorelbine is very similar to vinblastine in molecular formula, and is available in China. From November 2016 to March 2017, two patients with recurrent ALCL were recruited in the Department of Hematology and Oncology, Shanghai Children's Medical Center. They received vinorelbine monotherapy and achieved clinical remission (PET CR) at 8 weeks. One patient with bone marrow recurrence showed negative ALK / NPM by PCR . Based on this, the investigators will expand the sample to further investigate the therapeutic efficiency and safety of vinorelbine in children and adolescents with ALCL.

ELIGIBILITY:
Inclusion Criteria:

Children and adolescents with a clear diagnosis of recurrent / progressive ALCL at Shanghai Children's Medical Center or other centers since September 2017 include:

* Diagnosed as ALCL, already received first-line treatment, but get disease progression;
* After receiving ALCL treatment has got CR then diagnosed relapse, need for pathological diagnosis.

Exclusion Criteria:

* Patients with other systemic diseases, severe infections or critically illness.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2022-07 (Actual); Study Completion 2022-07 (Actual)

PRIMARY OUTCOMES:
Event free survival | 5 years

SECONDARY OUTCOMES:
Overall survival | 5 years

OTHER OUTCOMES:
Safety statistics: adverse reactions during the trial through NCI CTCAE version 4.0. | 2 years
  The investigators will record the adverse reactions during the trial through NCI CTCAE version 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Yijin Gao, MD, Principal Investigator — Shanghai Children's Medical Center
Locations (1):
- Shanghai Children's Medical Center, Shanghai, Shanghai Municipality, China